CLINICAL TRIAL: NCT05288790
Title: Microbiome Metabolites and Alcohol in HIV to Reduce CVD RCT
Acronym: META HIV CVD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: University of Louisville (Other); Boston University (Other)
Responsible Party: Principal Investigator, Matthew S.Freiberg, Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P01AA029542 (NIH)
Record Dates: First submitted 2022-02-28; First posted 2022-03-21 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Microtia; Dysbiosis; Alcohol Drinking; HIV Infections; Cardiovascular Diseases
MeSH Terms: conditions — Congenital Microtia; Dysbiosis; Alcohol Drinking; HIV Infections; Cardiovascular Diseases | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: This is a two-arm randomized double blind clinical trial study design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Supplement (Experimental): Probiotic
  Interventions: Dietary Supplement: Probiotic
- Study placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Dietary supplement
  Arms: Study Supplement
Dietary Supplement: Placebo — Placebo sachet
  Arms: Study placebo

SUMMARY:
Among people living with HIV, heavy drinking increases the risk of heart disease and death. Studies suggest that alcohol changes the number and kind of bacteria in your gut and these changes increase the risk of heart disease and death. This randomized controlled trial will determine whether a pill containing healthy gut bacteria can increase the number good bacteria in the gut, lower levels of inflammation, and lower the risk of heart disease and death.

DETAILED DESCRIPTION:
Among people living with HIV (PLWH), heavy drinking increases the risk of cardiovascular disease (CVD) and death. Data suggest that alcohol-associated gut dysbiosis partially drives this risk. Whether interventions targeting alcohol-associated gut dysbiosis among PLWH improve dysbiosis, lower levels of microbial translocation, inflammation, and harmful metabolites (e.g., trimethylamine N-oxide [TMAO)]) is unknown. The investigators' hypothesis for this P01 application is that among PLWH, a probiotic can mitigate or reduce alcohol associated gut dysbiosis and lower levels of microbial translocation, inflammation, and improve metabolite profiles (Project 1); and that harmful levels of these metabolites will be associated with higher CVD and death risk (Project 2). This team, with expertise in alcohol, HIV, gut microbiome, and biomarker research has conducted two NIAAA funded trials, a metabolite study, and a gut microbiome study among Russian PLWH who are heavy drinkers. Data from these studies show that among PLWH: (1) heavy drinking is associated with incident CVD, death and gut dysbiosis (characterized by a reduction in butyrate producing bacteria); and (2) this gut dysbiosis is associated with inflammation, altered bile acids, and high TMAO levels. Given these data and reports from pilot studies showing that probiotics are safe, may improve gut dysbiosis and reduce inflammation among PLWH, the investigators propose an RCT among 250 PLWH with heavy alcohol consumption who are on antiretroviral therapy and have CD4+ counts≥350 cells/mm3 to compare the effects of a probiotic tailored to alcohol associated gut dysbiosis vs. placebo to: (1) improve GI dysbiosis; (2) reduce plasma metabolite (e.g., TMAO) and biomarker levels of microbial translocation and inflammation; and (3) lower CVD and mortality risk. All participants will receive evidenced-based counseling for alcohol use. The specific aims will compare the effects of a tailored probiotic vs. placebo at 6 months on (Aim 1) dysbiosis (fecal Firmicutes to Bacteroidetes (F/B) ratio, primary study outcome; fecal Lachnospiraceae-family of butyrate producers) and plasma metabolites (plasma butyrate, deoxycholic acid:cholic acid ratio, and TMAO) (Aim 2) biomarkers of inflammation plasma, IL-6, D-dimer, sCD14), microbial translocation [Lipopolysaccharide binding protein], (Aim 3) cardiovascular risk (Reynolds risk score), mortality risk (VACS index); (Aim 4 exploratory) alcohol consumption (% heavy drinking days in past month) and HIV disease progression (CD4 cell count). The investigators hypothesize that as compared with placebo, the probiotic arm will have significantly: (1) higher F/B ratio and levels of fecal Lachnospiraceae, plasma butyrate, deoxycholic acid: cholic acid ratio and lower levels of TMAO; (2) lower plasma biomarker levels of microbial translocation and inflammation; (3) lower Reynolds risk score and VACS index; (4) lower % heavy drinking days in the past month and higher CD4 cell counts. The findings from this RCT, Microbiome, mETabolites, and Alcohol in HIV to reduce CVD (META HIV CVD RCT), will inform probiotics' role as standard adjunctive therapy complementing alcohol interventions among PLWH who are heavy drinkers.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected

Exclusion Criteria:

* Not fluent in English

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2026-08-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Firmicutes to Bacteroidetes ratio | 6 months
  Dysbiosis

SECONDARY OUTCOMES:
Intestinal permeability | 6, 12 months
  measuring levels of butyrate, deoxycholic acid:cholic acid ratio, and TMAO
Firmicutes to Bacteroidetes ratio | 12 months
  Dysbiosis measurement
Microbial Translocation | 6, 12 months
  measuring plasma lipopolysaccharide binding protein
Inflammation | 6, 12 months
  measuring plasma for interleukin 6 [IL-6], D-dimer, and sCD14

OTHER OUTCOMES:
Mortality | 6 and 12 months
  Veterans Aging Cohort Study Index Score (lower scores are better and higher scores are worse) (ranges from 0-164)
CVD risk | 6 and 12 months
  Reynolds Risk Score (the higher the score the higher the risk) (ranges from 100-400 mg/dL)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States